CLINICAL TRIAL: NCT04861948
Title: Phase Ib Study to Evaluate the Efficacy, Safety and Tolerability of IBI188 Combination Therapy in Subjects With Advanced Malignancies
Brief Title: IBI188 Combination Therapy in Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No signs of efficacy in solid tumors
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI188A104
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Solid Tumors; Lung Adenocarcinoma; Osteosarcoma
MeSH Terms: conditions — Adenocarcinoma of Lung; Osteosarcoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Cisplatin; Carboplatin; Bevacizumab; sintilimab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A (Experimental)
  Interventions: Drug: IBI188; Drug: Sintilimab
- Cohort B (Experimental)
  Interventions: Drug: IBI188; Drug: Cisplatin/Carboplatin; Drug: Bevacizumab; Drug: Pemetrexed
- Cohort C (Experimental)
  Interventions: Drug: IBI188; Drug: GM-CSF
- Cohort D (Experimental)
  Interventions: Drug: IBI188; Drug: Sintilimab

INTERVENTIONS:
Drug: IBI188 — intravenous
Drug: GM-CSF — subcutaneous injection
  Arms: Cohort C
Drug: Cisplatin/Carboplatin — intravenous
  Arms: Cohort B
Drug: Bevacizumab — intravenous
  Arms: Cohort B
Drug: Sintilimab — intravenous
  Arms: Cohort A; Cohort D
Drug: Pemetrexed — intravenous
  Arms: Cohort B

SUMMARY:
A Phase Ib study aim to evaluate the efficacy, safety, and tolerability of IBI188 combination therapy in subjects with advanced malignancies

ELIGIBILITY:
Inclusion Criteria:

1. Patients with locally advanced or metastatic solid tumors cannot be cured by surgery or other local treatments .
2. Aged ≥ 18 years (≥ 12 years is acceptable in Cohort C).
3. Able to provide archived or fresh tumor tissue samples for biomarker assessment.
4. Have at least one measurable lesion according to RECIST version 1.1.
5. ECCG PS score of 0-2.
6. Adequate organ and bone marrow functions .
7. Life expectancy ≥ 12 weeks.
8. Female subjects of childbearing potential or male subjects with partners of childbearing potential should take effective contraceptive measures throughout the whole treatment period and until 6 months after treatment.
9. Must voluntarily sign the Informed Consent Form (ICF), and be able to follow all study requirements and procedures. For the subjects enrolled in Cohort C who are ≥ 12 and < 18 years old, in addition to obtaining the child's own consent, their guardians should provide informed consent and sign the ICF.

Exclusion Criteria:

1. Previous exposure to any CD47 antibody, SIRPα antibody, CD47/SIRPα recombinant protein or other inhibitors that act in the same pathway.
2. Previous exposure to any anti-programmed death receptor 1 (PD-1) or anti-programmed death-ligand (PD-L1) antibody (except Cohort C).
3. Concurrent participation in another clinical study.
4. The last dose of anti-tumor therapy is within 4 weeks before the first dose of study treatment.
5. Have undergone major surgical procedures within 4 weeks prior to the first dose of study treatment or planned to receive major surgery during the study treatment.
6. Presence of toxicities (excluding alopecia and fatigue) induced by previous anti-tumor therapy that has not recovered to Grade 0 or 1 as assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 prior to the first dose of study treatment.
7. Known hypersensitivity to IBI188 or any ingredient in the study drug product.
8. History of other primary malignancies.
9. Female subjects who are pregnant or lactating.
10. Other ineligible conditions considered by the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 24 months
Adverse Events | 24 months
  Incidence, correlation with the study drug and severity of all adverse events (AEs), treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Progression-free survival | 24 months
Overall survival | 24 months
Disease control rate | 24 months
Duration of response | 24 months
Time to response | 24 months
Area Under Curve, AUC | 24 months
maximum concentration (Cmax) | 24 months
minimum concentration (Cmin) | 24 months
clearance (CL) | 24 months
volume of distribution (V) | 24 months
half-life (t1/2) | 24 months
Positive rate of anti-drug antibody (ADA) | 24 months
Positive rate of neutralizing antibody (NAb) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ba Yi, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital; Zhang Dahong, Principal Investigator — Zhejiang Provincial People's Hospital; Guo Hongqian, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Fang Meiyu, Principal Investigator — Zhejiang Cancer Hospital; Xie Yu, Principal Investigator — Hunan Cancer Hospital; Liu Jisheng, Principal Investigator — First Affiliated Hospital of Soochow University; Wang Ying, Principal Investigator — Zhejiang Provincial People's Hospital; Wang Haiying, Principal Investigator — Shougang Hospital, Peking University; Wang Mengzhao, Principal Investigator — Shougang Hospital, Peking University; Lv Qiang, Principal Investigator — Jiangsu Provincial People's Hospital; Li Xiangping, Principal Investigator — Nanfang Hospital, Southern Medical University; Liu Guihong, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University; Mou Weiqi, Principal Investigator — Chongqing University Cancer Hospital; Guo Wei, Principal Investigator — Peking Union Medical College; Wang Wei, Principal Investigator — Hunan Cancer Hospital; Xu Chongyuan, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China